CLINICAL TRIAL: NCT00197379
Title: The Study for New Effect of Roxithromycin on Androgenetic Alopecia.
Brief Title: The Effect of 0.5% Roxithromycin Lotion for Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamamatsu University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-61
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2005-04

CONDITIONS: Alopecia
Keywords: androgenetic alopecia; roxitromycin; apoptosis
MeSH Terms: conditions — Alopecia | interventions — Roxithromycin

INTERVENTIONS:
Drug: roxithromycin

SUMMARY:
The purpose of this study is exploiting the new drugs for androgenetic alopecia because there are still no effective and safe topical drug for androgenetic alopecia. Roxithomycin is one of the macrolide antibiotics that has immunomodulatory effects. We firstly found that roxithromycin increases the rate of murine and human hair follicle elongation in vitro. Therefore, we apply this drug on this disease therapy.

DETAILED DESCRIPTION:
The topical therapy for androgenetic alopecia is still not enough to improve cosmetically. Thereforem we try to find new effective and safe topical therapy for this disease. Roxithromycin has not only antibacterial action but also immunomodulatory and anti-inflamatory potency. For example, roxitromycin inhibits T cell responces to mitogens and production of cytokines, IL-2 and IL-5. We firstly found that roxitromycin increased human and murine hair elongation in vitro to inhibit apoptosis of hair bulb. Then, we wish to apply roxithromycin on the therapy for androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Androgenetic alopecia

Exclusion Criteria:

* Cicatricial alopecia
* Allergy to roxitromycin
* Children (19years old or younger)
* Pregnant female

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-05; Study Completion 2007-01 (Estimated)

SECONDARY OUTCOMES:
Pathological study taken from lesional scalp skin. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Takigawa, M.D., Study Chair — Hamamatsu University
Locations (1):
- Department of Dermatology, Hamamatsu University School of Medicine, Hamamatsu, Japan

REFERENCES:
- [Background] Ohshima A, Tokura Y, Wakita H, Furukawa F, Takigawa M. Roxithromycin down-modulates antigen-presenting and interleukin-1 beta-producing abilities of murine Langerhans cells. J Dermatol Sci. 1998 Jul;17(3):214-22. doi: 10.1016/s0923-1811(98)00017-6. PMID 9697050
- [Background] Ito T, Ito N, Saathoff M, Bettermann A, Takigawa M, Paus R. Interferon-gamma is a potent inducer of catagen-like changes in cultured human anagen hair follicles. Br J Dermatol. 2005 Apr;152(4):623-31. doi: 10.1111/j.1365-2133.2005.06453.x. PMID 15840090
- [Background] Lindner G, Botchkarev VA, Botchkareva NV, Ling G, van der Veen C, Paus R. Analysis of apoptosis during hair follicle regression (catagen). Am J Pathol. 1997 Dec;151(6):1601-17. PMID 9403711
- See also: Hamamatsu University School of Medicine — http://www.hama-med.ac.jp/